CLINICAL TRIAL: NCT04069676
Title: Emotional Proactive Brain Study in Adults With Autism Spectrum Condition
Acronym: PREDEMAUT
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.131; 2019-A01145-52 (Other: ID RCB)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Condition; predictive coding; visual perception; electroencephalography; autonomous nervous system; heart rate variability; electrodermal reactivity
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Condition (ASC): Adults males and females with a formal autism diagnosis, without intellectual disability
  Interventions: Other: EEG
- Typically developped (TD): Adults males and females without any neurodevelopemental issue (or health issue which could impaired task performances)
  Interventions: Other: EEG

INTERVENTIONS:
Other: EEG — EEG, ECG and EDR record during a behavioral task
  Other Names: ECG; EDR

SUMMARY:
This project aims:

* to study behavioral and cerebral activity specificity (latency and amplitude of evoked potentials, time frequency maps and cerebral connectivity) in predictive process (top-down regulation) during visual recognition of static and dynamic stimuli in adults participants with autism spectrum conditions compared to typically developed participants.
* to study the relation between predictive process and autonomous response (heart activity and electrodermal activity)
* to explore potential sex differences between autistic males and females

DETAILED DESCRIPTION:
Once eligibility criteria would have been verified, information on the study will be given and non opposition of the participant will be collected.Then, the participant will be comfortably installed in order to pass the Landolt C task (visual acuity task) on a computer. If his vision is normal, electroencephalogram (EEG), electrocardiogram (ECG) and electrodermal activity (EDA) of participants, will be recorded during visual processing and recognition tasks. Stimuli will include emotional and non emotional pictures and films, filtered in coarse-to-fine versus fine-to-coarse sequences in order to stimulate or not predictive process described by Bar (2007).

The participant will also have to complete an abbreviated version of the Wechsler Adult Intelligence Scale, IVth edition (Wechsler, 2003), and the Autism Spectrum Quotient (Baron-Cohen et al., 2001) if he never did it before. The aim is to pair as much as possible group by IQ and to verify that control participants don't present autistic traits above the Autism Spectrum Quotient cutoff. Groups will also be paired by age and education level.

ELIGIBILITY:
Inclusion Criteria:

* affiliation to the french social protection care
* information and non opposition of the participant
* information and non opposition of tutor/curator if the case presented
* normal or corrected to normal vision
* capacity to understand and apply instruction required by the task
* no participation in another research
* for autistic person: formal diagnosis of autism spectrum condition (autism/asperger/PDD-NS) according to CIM-10/DSM-IV/DSM-5 criteria

Exclusion Criteria:

* adults with no ability to express their consent
* adults on judiciary protection
* perceptive/motor/neurological/psychiatric issue
* major health issue (cardiac, metabolic ...)
* alcohol or drug consumption

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults autistic males and females without intellectual disability compared to a control group
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Differences between autistic and typically developed participants in evoked potentials related to prediction mechanisms during visual processing | 55 minutes recording
  - differences in evoked potentials (latency and amplitude) Changes will be assessed between coarse-to-fine and fine-to-coarse sequencies. It will be used to investigated how predictive mechanism during visual perception are affected in autism regarding cerebral activity.
Differences between autistic and typically developed participants in behavioral responses related to prediction mechanisms during visual processing | 55 minutes (same recording as before)
  - differences in behavioral responses (reaction time and correct response rate) Changes will be assessed between coarse-to-fine and fine-to-coarse sequencies. It will be used to investigated how predictive mechanism during visual perception are affected in autism regarding behavioral response.

SECONDARY OUTCOMES:
Differences between groups in oscillatory activity | 55 minutes (same record as before)
  -differences in time-frequency maps. Changes will be assessed between coarse-to-fine and fine-to-coarse sequencies. It will be used to investigated how predictive mechanism during visual perception are affected in autism regarding cerebral activity.
Difference between groups in cerebral connectivity | 55 minutes (same record as before)
  - differences in Dynamic Causal Modeling Changes will be assessed between coarse-to-fine and fine-to-coarse sequencies. It will be used to investigated how predictive mechanism during visual perception are affected in autism regarding cerebral activity.
Differences between groups in autonomous activity | 55 minutes (same record as before)
  * ECG activity (HRV analysis)
  * electrodermal activity (EDA) Changes will be assessed between coarse-to-fine and fine-to-coarse sequencies. It will be used to investigated how predictive mechanism during visual perception are affected in autism regarding autonomous activity.
Sex differences | 55 minutes (same record as before)
  - sex differences analysis Changes will be assessed between coarse-to-fine and fine-to-coarse sequencies. It will be used to investigated the existence of sex differences in autism regarding predictive process during visual perception.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Vercueil, Doctor, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

REFERENCES:
- [Background] Bar M. The proactive brain: using analogies and associations to generate predictions. Trends Cogn Sci. 2007 Jul;11(7):280-9. doi: 10.1016/j.tics.2007.05.005. Epub 2007 Jun 4. PMID 17548232
- [Background] Caplette L, Wicker B, Gosselin F. Atypical Time Course of Object Recognition in Autism Spectrum Disorder. Sci Rep. 2016 Oct 18;6:35494. doi: 10.1038/srep35494. PMID 27752088
- [Background] Gomot M, Wicker B. A challenging, unpredictable world for people with autism spectrum disorder. Int J Psychophysiol. 2012 Feb;83(2):240-7. doi: 10.1016/j.ijpsycho.2011.09.017. Epub 2011 Oct 1. PMID 21968196
- [Background] Peyrin C, Michel CM, Schwartz S, Thut G, Seghier M, Landis T, Marendaz C, Vuilleumier P. The neural substrates and timing of top-down processes during coarse-to-fine categorization of visual scenes: a combined fMRI and ERP study. J Cogn Neurosci. 2010 Dec;22(12):2768-80. doi: 10.1162/jocn.2010.21424. PMID 20044901
- [Background] Quintana DS, Guastella AJ, Outhred T, Hickie IB, Kemp AH. Heart rate variability is associated with emotion recognition: direct evidence for a relationship between the autonomic nervous system and social cognition. Int J Psychophysiol. 2012 Nov;86(2):168-72. doi: 10.1016/j.ijpsycho.2012.08.012. Epub 2012 Aug 30. PMID 22940643
- [Background] Sinha P, Kjelgaard MM, Gandhi TK, Tsourides K, Cardinaux AL, Pantazis D, Diamond SP, Held RM. Autism as a disorder of prediction. Proc Natl Acad Sci U S A. 2014 Oct 21;111(42):15220-5. doi: 10.1073/pnas.1416797111. Epub 2014 Oct 6. PMID 25288765
- [Background] Thayer JF, Ahs F, Fredrikson M, Sollers JJ 3rd, Wager TD. A meta-analysis of heart rate variability and neuroimaging studies: implications for heart rate variability as a marker of stress and health. Neurosci Biobehav Rev. 2012 Feb;36(2):747-56. doi: 10.1016/j.neubiorev.2011.11.009. Epub 2011 Dec 8. PMID 22178086